CLINICAL TRIAL: NCT03722017
Title: Drug Reduction in Older Patients: The DROP Trial
Acronym: DROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 17-033
Record Dates: First submitted 2018-10-09; First posted 2018-10-26 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Geriatric Assessment; Frail Elderly; Skilled Nursing Facilities; Patient-centered Care
Keywords: deprescriptions; polypharmacy; potentially inappropriate medication; medication adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: The investigators will ascertain for each medication: (1) Indication; (2) Deprescribing rationale (i.e., stopping or reducing dose) for each medication.
  Deprescribing Recommendations will be specified as: (1) Stop prior to hospital discharge, no monitoring; (2) Stop prior to hospital discharge with monitoring; (3) Stop at specified time point following hospital discharge; (4) Reduce over time with monitoring until stopped; (5) Reduce to lower dose without monitoring; (6) Reduce to lower dose with monitoring. Deprescribing will begin prior to hospital discharge.
  The investigators will incorporate Veteran preferences, communicate with all providers involved in prescribing, create final deprescribing actions, and do enhanced hospital discharge communication.
Masking Description: The participant and providers involved in their care will not be masked to the intervention, as there is participation of both groups in the deprescribing protocol discussions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control--usual care (No Intervention): Medication History: All participants / surrogates will receive a structured interview and chart review by the study Pharmacist or Nurse Practitioner at enrollment to determine:
  Medications: Medications will include ANY medication with the potential for continuation at the time of hospital discharge to include pre-hospital medications, [OTC medications] and active in-hospital medications. Pre-hospital [and OTC] medications will be confirmed by Veteran/surrogate interview and pharmacy refills. If a Veteran is admitted from SNF (short-term stay), the investigators will request a copy of the Medication Administration Record (MAR) for the past 30 days. Current medications will be defined as those taken within 30 days prior to the index (enrollment) hospitalization event.
- Intervention--deprescribing protocol (Experimental): In addition to a medication history, a study Pharmacist or Nurse Practitioner will review the reconciled total enrollment medication list. The following information will be ascertained for each medication: (1) Medication Indication; and, (2) Deprescribing rationale: Rationales for deprescribing (i.e., stopping or reducing dose) will be assessed for each medication.
  Deprescribing Recommendations: For each medication recommended for deprescribing, the deprescribing action will be specified as: (1) Stop prior to hospital discharge without need for monitoring; (2) Stop prior to hospital discharge with symptoms/physiologic monitoring; (3) Stop at specified time point following hospital discharge; (4) Reduce over time with monitoring until medication is stopped; (5) Reduce to lower dose without need for monitoring; (6) Reduce to lower dose with symptoms/physiologic monitoring.
  Interventions: Other: Deprescribing intervention

INTERVENTIONS:
Other: Deprescribing intervention — In addition to a medication history, a study Pharmacist or Nurse Practitioner will review the reconciled total enrollment medication list. The following information will be ascertained for each medication: (1) Medication Indication; and, (2) Deprescribing rationale: Rationales for deprescribing (i.e., stopping or reducing dose) will be assessed for each medication.
  Deprescribing Recommendations: For each medication recommended for deprescribing, the deprescribing action will be specified as: (1) Stop prior to hospital discharge without need for monitoring; (2) Stop prior to hospital discharge with symptoms/physiologic monitoring; (3) Stop at specified time point following hospital discharge; (4) Reduce over time with monitoring until medication is stopped; (5) Reduce to lower dose without need for monitoring; (6) Reduce to lower dose with symptoms/physiologic monitoring.
  Arms: Intervention--deprescribing protocol

SUMMARY:
Project Objectives: The proposed randomized, controlled trial will evaluate the effects of procedures to reduce medications among hospitalized older Veterans discharged to nursing homes using an hybrid study design to inform future efforts to spread it across VA.

Project Background/Rationale: Patients discharged to nursing homes for short stays represent the largest group of Medicare beneficiaries discharged to post-hospital services and are a particularly high risk group for loss of independence and other poor clinical outcomes. This investigative team recently completed a VA-funded Quality Improvement Award and a Centers for Medicare and Medicaid Services (CMS) Innovation Award, both of which provide strong results related to the occurrence of polypharmacy and the relationship between polypharmacy and geriatric syndromes (e.g., medications associated with falls) in this patient population. Based on these data, the investigators developed and pilot-tested a patient-centered deprescribing set of procedures combined with standardized questions for eight geriatric syndromes to be implemented in the hospital and monitored during the nursing home stay.

Project Methods: The investigators propose an innovative hybrid study design that will be conducted in one VA hospital. The goal of the proposed DROP intervention is to safely deprescribe medications, as defined by reducing doses or stopping medications, based on a combination of clinical criteria and Veteran preferences. This randomized, controlled trial conducted over three years will evaluate the effects of this hospital-based intervention on medication use, geriatric syndromes, and health status across Veterans' care transitions from the hospital to nursing home to home to include a 90-day follow-up period after leaving the nursing home. The hypothesis is that reducing medications for older Veterans will favorably impact geriatric syndromes. Additionally, the investigators aim to understand Veteran, both VA and non-VA provider and system-level factors that help or hinder how well the deprescribing procedures are implemented to inform future clinical uptake and dissemination throughout the VA.

DETAILED DESCRIPTION:
Overview and Specific Aims Polypharmacy, defined as five or more medications, is common in older patients discharged to skilled nursing facilities (SNFs) and is associated with adverse health outcomes. As part of a recent VA project, the investigators prospectively collected medication data for 134 hospitalized, older Veterans. These data showed that, on average, 14.2 medications were ordered for Veterans discharged to SNF, which included 2.5 medications newly prescribed in the hospital that met criteria for being potentially inappropriate medications (PIMs). Moreover, 75% of these Veterans had two or more geriatric syndromes. Geriatric syndromes are clinical conditions common in older adults such as cognitive impairment, unintentional weight loss and falls. The co-occurrence of multiple syndromes is associated with loss of independence and higher healthcare utilization. All Veterans with polypharmacy also had one or more medications associated with geriatric syndromes. The prevalence of polypharmacy and multiple geriatric syndromes may partially explain why these patients often have poor health outcomes after SNF discharge. Recent data suggests that only 28% of patients discharged from SNF are living at home 100 days later, and 35% experience an adverse drug event.

There is a dearth of evidence related to the management of multiple co-existing geriatric syndromes, and few interventions have been implemented to reduce medications while also monitoring health outcomes. The relationship between polypharmacy, adverse drug events and geriatric syndromes in the VA population supports the rationale for an intervention focused on deprescribing medications before hospital discharge. The investigators have pilot-tested a multifaceted intervention (Drug Reduction in Older Patients, DROP) to engage patients and providers to reduce the number and/or dose of medications prior to hospital discharge. The proposed randomized, controlled trial is powered to evaluate the effect of this intervention on a reduction in medications as defined by the total number of prescribed medications, the number of PIMs, anticholinergic and sedative drug burden and the number of medications associated with geriatric syndromes. In addition, the investigators will collect relevant data on the prevalence and severity of geriatric syndromes and other clinical outcomes. The investigators also will use a hybrid research design to evaluate both effectiveness and implementation issues to better inform future adoption and sustainability. Our overarching hypothesis is that a hospital-based intervention to safely reduce the total number of medications represents the most feasible way to impact multiple health-related outcomes among older Veterans. Our Specific Aims reflect the primary outcomes that are the focus of the analyses, although the investigators also will measure secondary outcomes related to VA healthcare utilization and patient safety:

Specific Aim 1: Implement a patient-centered deprescribing intervention (DROP) in the hospital to reduce the total number of medications Veterans are prescribed at hospital discharge.

Specific Aim 2: Document the effects of a Veteran-centered deprescribing intervention (DROP) on medication adherence, health status, and geriatric syndromes.

Specific Aim 3: Evaluate intervention implementation to inform future adoption and sustainability.

Potential for Impact: The DROP intervention has significant potential to impact the health of older hospitalized Veterans vulnerable to poor health outcomes. During hospitalization and SNF care, older Veterans often acquire new geriatric syndromes and medications, exactly when deprescribing actions should be initiated by care providers in the context of clinical oversight. Lastly, the application of an innovative hybrid research design will allow us to collect critical data related to both intervention effectiveness and implementation to better inform future adoption and sustainability across the VA.

Innovation: Our study is advancing science in multiple ways:

1. The proposed study reflects one of the first controlled intervention trials designed to improve post discharge outcomes for the high-risk population of older Veterans transitioning from hospital to SNF to home. Healthcare costs are increasing for this patient population, and they are at high risk for medication-associated complications and newly acquired geriatric syndromes.
2. Although the number of medications is strongly associated with increases in geriatric syndromes, it is unknown whether reducing medications will improve geriatric syndromes. This trial will generate data to evaluate the impact of medication reduction on Veteran health outcomes.
3. To date, there have been no controlled intervention trials focused on reducing the number of medications prescribed for hospitalized patients discharged to SNF, and the proposed intervention is one of the first to explicitly incorporate Veteran preferences into deprescribing efforts, which is consistent with Veteran-centered care initiatives. Moreover, our preliminary data show that incorporating patient preferences in the intervention protocol significantly changes these clinical decisions.
4. The proposed trial will evaluate both clinical effectiveness and implementation to inform the potential for DROP to be adopted into VA clinical practice.

Rationale for VA Study: Dr. Simmons was recently awarded an National Institute on Aging (NIA) R01 focused on polypharmacy in hospitalized non-Veterans. The investigators summarize below the primary differences between the two studies and our rationale for the importance of the proposed VA study:

The Need for More Evidence: Our NIA study focuses on non-Veterans hospitalized at Vanderbilt University Medical Center (VUMC) and discharged to a select group of SNFs that have partnered with VUMC for post-acute care services. Unfortunately, the scope of the NIA study does not allow us to evaluate the intervention in two separate healthcare systems with two unique patient populations and a larger number of SNFs, to include VA Community Living Centers and VA contract community nursing homes.

Uniqueness of the Veteran population: Our preliminary data demonstrates important differences in older hospitalized Veterans and non-Veterans discharged to SNF. Beyond being predominately male, older Veterans in the investigators' prior study had a higher overall prevalence of geriatrics syndromes and were prescribed more medications at hospital discharge than non-Veterans, particularly antidepressants and antipsychotics. Data also suggests that Veterans may be more willing to reduce their medicines; thus, the magnitude of the intervention effects may differ in the VA. Finally, hospitalized Veterans are discharged to a diverse group of SNFs, many of which are located in rural communities. Unlike the investigators' NIA study, which only includes a select group of partner SNFs predominately located in an urban area close to Vanderbilt, the proposed study will follow Veterans from hospital to SNF to home, irrespective of which SNF they utilize. The VA study, therefore, will more closely mimic real-world practice. The innovative application of an effectiveness-implementation hybrid design will further inform unique aspects of the VA healthcare system critical to adoption.

Uniqueness of VA healthcare system: The VA healthcare system differs significantly from other hospital systems, to include medication prescribing practices and how patients access and pay for medications. Thus, the investigators do not expect the results of the NIA study at VUMC to be directly translatable into the VA healthcare system. The proposed study also will yield an understanding of Veteran and VA provider attitudes toward deprescribing and other system factors unique to the VA that may influence intervention implementation.

Note: The investigators resumed face to face enrollment for non-COVID patients as of 8/17/20. COVID+ patients were being approached by phone.

Note: Investigators focus the reporting on primary medication outcomes for two reasons: (1) to align with reporting of an NIH/NIA funded deprescribing trial that utilized a near identical intervention (NCT02979353); and (2) medication outcomes had the strongest statistical power. Variable response rates across multiple timepoints for Veteran-reported secondary outcome measures limited the statistical power to detect intervention effects on secondary outcomes. Additionally, results for the 7-day post-SNF follow up timepoint are not presented due to a protocol change mid-study that resulted in incomplete data for that timepoint. The protocol change allowed the study to retain Veterans who were referred to a SNF but ultimately discharged directly home from the hospital (instead of SNF); thus, a significant proportion of enrolled Veterans have no data for the 7-day post-SNF follow up.

ELIGIBILITY:
Inclusion Criteria:

* Referred to SNF (per Physical Therapy and/or Social Work notes)
* Being discharged from the Nashville VA hospital from a medicine or orthopedics team
* Age > or = 50
* Have polypharmacy, as defined by > 5 medications based on pre-hospital and in-hospital medications
* Able to self-consent or has a surrogate

Exclusion Criteria:

* Resides in long-term care
* On hospice
* Not expected to discharge within 48 hours of referral

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Mixon, MD MSPH MS, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share our protocol and a de-identified anonymized dataset.
Supporting Information: Study Protocol
Time Frame: Data will become available Oct 31, 2021 (study conclusion).
Access Criteria: A de-identified dataset will be shared upon the finalization of a written agreement between VA Tennessee Valley Healthcare System and the requesting party. This agreement will detail use of the data and prohibit the re-identification of dataset subjects. Our study team will evaluate requests for datasets.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at the Nashville VA Medical Center (part of the Tennessee Valley VA Health Services) from October 2019 through November 2022. A total of 260 veterans were enrolled.
Groups:
- Control--usual Care: Participants assigned to the control group will receive usual care as it is normally provided by the hospital and skilled nursing facility treatment teams. Research staff will monitor their prescribed medications in both care settings but not make any recommendations or changes, unless a safety issue is identified.
- Intervention--deprescribing Protocol: Participants assigned to the intervention group will receive a clinical review of their prescribed medications by a research clinician (Nurse Practitioner, Physician, or Pharmacist) followed by a patient interview to assess their willingness to deprescribe medications based on the study team's recommendations. The study team will coordinate with the participant's hospital treatment team to ensure the medication dose reductions or discontinuations to which the participant agreed were reflected in the hospital discharge orders. The goal of the intervention is to safely deprescribe medications based on both clinical criteria and Veteran preference.
Period: Overall Study
Arm/Group | Control--usual Care | Intervention--deprescribing Protocol
Started | 130 | 130
Hospital Discharge | 123 | 122
SNF Discharge | 70 | 84
7-Day Follow-Up | 99 | 104
Completed | 89 | 94
Not Completed | 41 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control--usual Care | Intervention--deprescribing Protocol | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  years
    number analyzed (Participants) | 129 | 130 | 259
    (all) | 72 [66 to 78] | 73 [66 to 77] | 72 [66 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  Participants
    number analyzed (Participants) | 129 | 130 | 259
    Female | 15 | 8 | 23
    Male | 114 | 122 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 123 | 124 | 247
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 29 | 51
  White | 105 | 94 | 199
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 130 | 260
Vulnerable Elders Survey 13 (VES-13) [Median (Inter-Quartile Range); unit: Score on a Scale] — The Vulnerable Elders Survey 13 (VES-13) is a self-rating of functional health status, and it consists of 4 groups of questions: age, self-perceived health, difficulties to perform 6 specific activities, and difficulties to perform daily living tasks due to health concerns. The total score ranges from 0 to 10. A score >=3 was considered to show impairment (i.e., worse outcome). Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  Score on a Scale
    number analyzed (Participants) | 111 | 115 | 226
    (all) | 6 [3 to 7] | 6 [3 to 7] | 6 [3 to 7]
Adherence to Refills and Medication Scale (ARMS) [Median (Inter-Quartile Range); unit: Score on a Scale] — Trained research staff administered the Adherence to Refills and Medication Scale (ARMS). Participants indicate the extent of their adherence on a 4-point Likert-like scale. Responses range from 1="none of the time" to 4="all of the time," and are summed to produce an overall adherence score ranging from 12-48, with lower values indicating better adherence (better outcome). Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  Score on a Scale
    number analyzed (Participants) | 93 | 94 | 187
    (all) | 15 [13 to 18] | 15 [13 to 17.8] | 15 [13 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Medications
Description: The number of medications a participant is taking. This includes all prescribed and over-the-counter medications and both scheduled and as-needed (PRN) medications.
Time Frame: Hospital Discharge, SNF Discharge, and 90-days after SNF Discharge
Population: Outcomes are reported for three different study time points (Hospital Discharge, Skilled Nursing Facility [SNF] Discharge, and 90-Day Follow Up After SNF Discharge). Both the Intervention and Control groups experienced attrition at each time point. The "number analyzed" below for each time point reflects the number of participants who completed that particular study time point.
Measure: Median (Inter-Quartile Range); unit: Medications
Arm/Group | Control--usual Care | Intervention--deprescribing Protocol
Number analyzed (Participants) | 123 | 122
Medications
  Hospital Discharge - approximately 5 days after enrollment | 15 [12 to 19] | 13 [11 to 17]
  SNF Discharge - approximately 30 days after enrollment: number analyzed (Participants) | 70 | 84
  SNF Discharge - approximately 30 days after enrollment | 15.5 [12 to 18] | 14 [10 to 17]
  90 Day Follow Up- approximately 110 days after enrollment: number analyzed (Participants) | 89 | 94
  90 Day Follow Up- approximately 110 days after enrollment | 15 [11 to 17] | 12.5 [10 to 16]
Statistical Analysis 1: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 1 applies to the Hospital Discharge Timepoint; Test type: Superiority; p = 0.006, Mixed Models Analysis; Risk Ratio (RR) = 0.91
Statistical Analysis 2: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 2 applies to the SNF Discharge Timepoint; Test type: Superiority; p = 0.110, Mixed Models Analysis; Risk Ratio (RR) = 0.93
Statistical Analysis 3: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 3 applies to the 90 Day Follow-Up Timepoint; Test type: Superiority; p = 0.060, Mixed Models Analysis; Risk Ratio (RR) = 0.92

2. Secondary Outcome: Total Drug Burden Index (DBI): Anticholinergic and Sedative Drug Burden
Description: A Drug Burden Index (DBI) score is calculated for each anticholinergic and sedative medication by dividing the individual medication's prescribed daily dose by the sum of the minimum effective dose (per FDA minimum recommended dose) and the patient's daily dose. The score range for each individual medication is 0 to 1, and the Anticholinergic & Sedative DBI reported is the sum of the individual medication scores. The Anticholinergic & Sedative DBI has a minimum score of 0 and no maximum. Higher scores indicate a higher drug burden (i.e., lower score is a better outcome).
Time Frame: Hospital Discharge, SNF Discharge, and 90 Days after SNF Discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control--usual Care | Intervention--deprescribing Protocol
Number analyzed (Participants) | 123 | 122
score on a scale
  Hospital Discharge - approximately 5 days after enrollment | 2.6 [1.6 to 3.7] | 2.6 [1.5 to 3.7]
  SNF Discharge - approximately 30 days after enrollment: number analyzed (Participants) | 70 | 84
  SNF Discharge - approximately 30 days after enrollment | 2.7 [1.5 to 3.9] | 2.6 [1.7 to 3.9]
  90 Day Follow Up- approximately 110 days after enrollment | 2.3 [1.2 to 3.4] | 2.2 [1.4 to 3.5]
Statistical Analysis 1: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 1 applies to the Hospital Discharge Timepoint; Test type: Superiority; p = 0.738, Mixed Models Analysis; Mean Difference (Net) = -0.049
Statistical Analysis 2: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 2 applies to the SNF Discharge Timepoint; Test type: Superiority; p = 0.995, Mixed Models Analysis; Mean Difference (Net) = 0.001
Statistical Analysis 3: Comparison: Control--usual Care vs Intervention--deprescribing Protocol; Statistical Analysis 3 applies to the 90 Day Follow Up Timepoint; Test type: Superiority; p = 0.721, Mixed Models Analysis; Mean Difference (Net) = 0.058

ADVERSE EVENTS:
Time Frame: Enrollment to 90-days post SNF Discharge (duration each participants' time in the study)
Description: Serious adverse events included escalation of care to the intensive care unit (during baseline hospitalization), rehospitalization (after baseline), and death.
Arm/Group | Control--usual Care | Intervention--deprescribing Protocol
All-Cause Mortality (participants affected / at risk) | 9/130 | 5/130
Serious Adverse Events (participants affected / at risk) | 57/130 | 60/130
Other Adverse Events (participants affected / at risk) | 13/130 | 14/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control--usual Care (N=130) | Intervention--deprescribing Protocol (N=130)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 3 (4)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmias (Cardiac disorders) | 5 (5) | 4 (4)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 3 (3)
Heart Failure (Cardiac disorders) | 7 (10) | 8 (10)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2)
Gastrointestinal motility and defecation condition (Gastrointestinal disorders) | 3 (4) | 2 (2)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 0 (0) | 1 (1)
General systems disorders (General disorders) | 2 (2) | 1 (1)
Alcoholic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 1 (5)
Bacterial infectious disorders (Infections and infestations) | 2 (2) | 1 (1)
Infections - pathogen unspecified (Infections and infestations) | 4 (4) | 8 (10)
Pneumonia (Infections and infestations) | 6 (7) | 5 (5)
Sepsis - pathogen unspecified (Infections and infestations) | 6 (7) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Viral infectious disoders (Infections and infestations) | 3 (3) | 4 (4) — COVID-19
Bone and joint fractures (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Procedural related injuries and complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Glucose metabolism disorder (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuro Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system vascular disorders (Nervous system disorders) | 4 (4) | 4 (4)
Neurotoxicity (Nervous system disorders) | 2 (2) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 3 (3)
Mental disorders (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal orientation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal disorders (Renal and urinary disorders) | 2 (2) | 4 (4)
Urinary tract signs and symptoms (Renal and urinary disorders) | 1 (1) | 1 (1)
Bronchial disorders (excludes neoplasms) (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Embolism and thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Failure to thrive (Social circumstances) | 1 (1) | 3 (3)
Hypothermia (Social circumstances) | 0 (0) | 1 (1)
Embolism and thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral edema (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
Vascular hypertensive disorders (Vascular disorders) | 1 (1) | 1 (1)
Vascular hypotensive disorders (Vascular disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control--usual Care (N=130) | Intervention--deprescribing Protocol (N=130)
Fall (Injury, poisoning and procedural complications) | 6 (9) | 6 (6)
Gastrointestinal motility and defecation condition (Gastrointestinal disorders) | 4 (4) | 4 (5)
Infections - pathogen unspecified (Infections and infestations) | 4 (4) | 2 (2)
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03722017/Prot_SAP_000.pdf